CLINICAL TRIAL: NCT00661453
Title: Phase I/II Trial of Valproic Acid and Carnitine in Infants With Spinal Muscular Atrophy Type I (CARNI-VAL Type I)
Brief Title: CARNIVAL Type I: Valproic Acid and Carnitine in Infants With Spinal Muscular Atrophy (SMA) Type I
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Families of Spinal Muscular Atrophy (Other); Leadiant Biosciences, Inc. (Industry)
Responsible Party: Principal Investigator, Kathryn Swoboda, Associate Professor, Neurology and Pediatrics Director, Pediatric Motor Disorders Research Program, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25409; IND 79276
Record Dates: First submitted 2008-04-14; First posted 2008-04-18 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Spinal Muscular Atrophy Type I
Keywords: Spinal Muscular Atrophy; SMA; Valproic Acid
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Atrophy, Spinal | interventions — Valproic Acid; Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All patients will receive VPA and carnitine.
  Interventions: Drug: Valproic Acid and Levocarnitine

INTERVENTIONS:
Drug: Valproic Acid and Levocarnitine — Drug: Valproic Acid and Levocarnitine; syrup; dosage is by weight

SUMMARY:
This is a multi-center trial to test safety and evaluate early treatment intervention with valproic acid and carnitine in moderating SMA symptoms of Type I infants.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a genetic disorder that results in severe muscle weakness. It is one of the most common conditions causing muscle weakness in children. Patients with SMA most often develop weakness as babies or young children. Most people with SMA gradually lose muscle strength and abilities over time. Babies with the severe infantile form of SMA, SMA type I, usually lose abilities and strength quickly over a few weeks or months.

Valproic acid (VPA) is a medicine that has been used for many years to treat patients with epilepsy. Recent research suggests that VPA may be able to upregulate expression of a backup copy of the SMN gene in SMA patient cell lines. In addition, some preliminary data suggests it may prolong survival in animal models of SMA. Because VPA can deplete carnitine in children with SMA Type I, carnitine is added to help prevent possible toxicity.

In this multi-center trial, we will evaluate the effects of VPA/carnitine on infants with SMA type I. A variety of outcome measures, including assessment of safety, will be performed at each study visit to follow the course of the disease. The protocol includes two baseline visits over a period of two weeks, two clinical assessments on medication at 3 and 6 months, and then 6 months additional followup via telephone. Total duration of the study will be approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory documentation of SMN mutation/deletion consistent with a genetic diagnosis of SMA
* Clinical diagnosis of SMA type I
* Age 2 weeks to 12 months
* Written informed consent of parents/guardian

Exclusion Criteria:

* Any clinical or laboratory evidence of hepatic or pancreatic insufficiency.
* Laboratory results drawn within 14 days prior to start of study drug demonstrating:

Liver transaminases (AST, ALT), lipase, amylase: > 1.5 x ULN White Blood Cell Count: < 3 Neutropenia: <1 Platelet: <100K Hematocrit: <30, persisting over a 30-day period

* Serious illness requiring systemic treatment and/or hospitalization within two weeks prior to study entry.
* Use of medications or supplements within 30 days of study enrollment that interfere with VPA or carnitine metabolism; that increase the potential risks of VPA or carnitine; or that are hypothesized to have a beneficial effect in SMA animal models or human neuromuscular disorders, including riluzole, valproic acid, hydroxyurea, oral use of albuterol, sodium phenylbutyrate, butyrate derivatives, creatinine, growth hormone, anabolic steroids, probenecid, oral or parenteral use of corticosteroids at entry, or agents anticipated to increase or decrease muscle strength or agents with presumed histone deacetylase (HDAC) inhibition.
* Infants who have participated in a treatment trial for SMA within 30 days of study entry or who will become enrollees in any other treatment trial during the course of this study.
* Unwillingness to travel for study assessments.
* Coexisting medical conditions that contradict use of VPA/carnitine or travel to and from study site.

Ages: 2 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Swoboda, M.D., Principal Investigator — University of Utah; Sandra P Reyna, M.D., Study Director — Families of Spinal Muscular Atrophy
Locations (8):
- United States (6):
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center, Dept. of Neurology, Columbus, Ohio
  - University of Utah/Primary Children's Medical Center, Salt Lake City, Utah
  - University of Wisconsin Children's Hospital, Madison, Wisconsin
- Hospital Sainte-Justine, Montreal, Quebec, Canada
- Klinikum der Universität zu Köln, Cologne, Germany

REFERENCES:
- [Background] Brahe C, Bertini E. Spinal muscular atrophies: recent insights and impact on molecular diagnosis. J Mol Med (Berl). 1996 Oct;74(10):555-62. doi: 10.1007/s001090050059. PMID 8912176
- [Background] Roberts DF, Chavez J, Court SD. The genetic component in child mortality. Arch Dis Child. 1970 Feb;45(239):33-8. doi: 10.1136/adc.45.239.33. PMID 4245389
- [Background] Pearn J. Incidence, prevalence, and gene frequency studies of chronic childhood spinal muscular atrophy. J Med Genet. 1978 Dec;15(6):409-13. doi: 10.1136/jmg.15.6.409. PMID 745211
- [Background] Czeizel A, Hamula J. A hungarian study on Werdnig-Hoffmann disease. J Med Genet. 1989 Dec;26(12):761-3. doi: 10.1136/jmg.26.12.761. PMID 2614795
- [Background] Emery AE. Population frequencies of inherited neuromuscular diseases--a world survey. Neuromuscul Disord. 1991;1(1):19-29. doi: 10.1016/0960-8966(91)90039-u. PMID 1822774
- [Background] Merlini L, Stagni SB, Marri E, Granata C. Epidemiology of neuromuscular disorders in the under-20 population in Bologna Province, Italy. Neuromuscul Disord. 1992;2(3):197-200. doi: 10.1016/0960-8966(92)90006-r. PMID 1483045
- [Background] Pearn J. Classification of spinal muscular atrophies. Lancet. 1980 Apr 26;1(8174):919-22. doi: 10.1016/s0140-6736(80)90847-8. PMID 6103267
- [Background] Bromberg MB, Swoboda KJ. Motor unit number estimation in infants and children with spinal muscular atrophy. Muscle Nerve. 2002 Mar;25(3):445-7. doi: 10.1002/mus.10050. PMID 11870724
- [Background] Swoboda KJ, Prior TW, Scott CB, McNaught TP, Wride MC, Reyna SP, Bromberg MB. Natural history of denervation in SMA: relation to age, SMN2 copy number, and function. Ann Neurol. 2005 May;57(5):704-12. doi: 10.1002/ana.20473. PMID 15852397
- [Background] Crawford TO. From enigmatic to problematic: the new molecular genetics of childhood spinal muscular atrophy. Neurology. 1996 Feb;46(2):335-40. doi: 10.1212/wnl.46.2.335. No abstract available. PMID 8614490
- [Background] Gilliam TC, Brzustowicz LM, Castilla LH, Lehner T, Penchaszadeh GK, Daniels RJ, Byth BC, Knowles J, Hislop JE, Shapira Y, et al. Genetic homogeneity between acute and chronic forms of spinal muscular atrophy. Nature. 1990 Jun 28;345(6278):823-5. doi: 10.1038/345823a0. PMID 1972783
- [Background] Melki J, Lefebvre S, Burglen L, Burlet P, Clermont O, Millasseau P, Reboullet S, Benichou B, Zeviani M, Le Paslier D, et al. De novo and inherited deletions of the 5q13 region in spinal muscular atrophies. Science. 1994 Jun 3;264(5164):1474-7. doi: 10.1126/science.7910982.
- [Background] Monani UR, Lorson CL, Parsons DW, Prior TW, Androphy EJ, Burghes AH, McPherson JD. A single nucleotide difference that alters splicing patterns distinguishes the SMA gene SMN1 from the copy gene SMN2. Hum Mol Genet. 1999 Jul;8(7):1177-83. doi: 10.1093/hmg/8.7.1177. PMID 10369862
- [Background] Campbell L, Potter A, Ignatius J, Dubowitz V, Davies K. Genomic variation and gene conversion in spinal muscular atrophy: implications for disease process and clinical phenotype. Am J Hum Genet. 1997 Jul;61(1):40-50. doi: 10.1086/513886. PMID 9245983
- [Background] Lefebvre S, Burlet P, Liu Q, Bertrandy S, Clermont O, Munnich A, Dreyfuss G, Melki J. Correlation between severity and SMN protein level in spinal muscular atrophy. Nat Genet. 1997 Jul;16(3):265-9. doi: 10.1038/ng0797-265. PMID 9207792
- [Background] Monani UR, Sendtner M, Coovert DD, Parsons DW, Andreassi C, Le TT, Jablonka S, Schrank B, Rossoll W, Prior TW, Morris GE, Burghes AH. The human centromeric survival motor neuron gene (SMN2) rescues embryonic lethality in Smn(-/-) mice and results in a mouse with spinal muscular atrophy. Hum Mol Genet. 2000 Feb 12;9(3):333-9. doi: 10.1093/hmg/9.3.333. PMID 10655541
- [Background] Feldkotter M, Schwarzer V, Wirth R, Wienker TF, Wirth B. Quantitative analyses of SMN1 and SMN2 based on real-time lightCycler PCR: fast and highly reliable carrier testing and prediction of severity of spinal muscular atrophy. Am J Hum Genet. 2002 Feb;70(2):358-68. doi: 10.1086/338627. Epub 2001 Dec 21. PMID 11791208
- [Background] Mailman MD, Heinz JW, Papp AC, Snyder PJ, Sedra MS, Wirth B, Burghes AH, Prior TW. Molecular analysis of spinal muscular atrophy and modification of the phenotype by SMN2. Genet Med. 2002 Jan-Feb;4(1):20-6. doi: 10.1097/00125817-200201000-00004. PMID 11839954
- [Background] Fischer U, Liu Q, Dreyfuss G. The SMN-SIP1 complex has an essential role in spliceosomal snRNP biogenesis. Cell. 1997 Sep 19;90(6):1023-9. doi: 10.1016/s0092-8674(00)80368-2. PMID 9323130
- [Background] Chang JG, Hsieh-Li HM, Jong YJ, Wang NM, Tsai CH, Li H. Treatment of spinal muscular atrophy by sodium butyrate. Proc Natl Acad Sci U S A. 2001 Aug 14;98(17):9808-13. doi: 10.1073/pnas.171105098. PMID 11504946
- [Background] Andreassi C, Jarecki J, Zhou J, Coovert DD, Monani UR, Chen X, Whitney M, Pollok B, Zhang M, Androphy E, Burghes AH. Aclarubicin treatment restores SMN levels to cells derived from type I spinal muscular atrophy patients. Hum Mol Genet. 2001 Nov 15;10(24):2841-9. doi: 10.1093/hmg/10.24.2841. PMID 11734549
- [Background] Brichta L, Hofmann Y, Hahnen E, Siebzehnrubl FA, Raschke H, Blumcke I, Eyupoglu IY, Wirth B. Valproic acid increases the SMN2 protein level: a well-known drug as a potential therapy for spinal muscular atrophy. Hum Mol Genet. 2003 Oct 1;12(19):2481-9. doi: 10.1093/hmg/ddg256. Epub 2003 Jul 29. PMID 12915451
- [Background] Andreassi C, Angelozzi C, Tiziano FD, Vitali T, De Vincenzi E, Boninsegna A, Villanova M, Bertini E, Pini A, Neri G, Brahe C. Phenylbutyrate increases SMN expression in vitro: relevance for treatment of spinal muscular atrophy. Eur J Hum Genet. 2004 Jan;12(1):59-65. doi: 10.1038/sj.ejhg.5201102. PMID 14560316
- [Background] Bohmer T, Rydning A, Solberg HE. Carnitine levels in human serum in health and disease. Clin Chim Acta. 1974 Nov 20;57(1):55-61. doi: 10.1016/0009-8981(74)90177-6. No abstract available. PMID 4279150
- [Background] Brooks H, Goldberg L, Holland R, Klein M, Sanzari N, DeFelice S. Carnitine-induced effects on cardiac and peripheral hemodynamics. J Clin Pharmacol. 1977 Oct;17(10 Pt 1):561-8. doi: 10.1177/009127007701701003. No abstract available. PMID 915022
- [Background] Christiansen RZ, Bremer J. Active transport of butyrobetaine and carnitine into isolated liver cells. Biochim Biophys Acta. 1976 Nov 2;448(4):562-77. doi: 10.1016/0005-2736(76)90110-3. PMID 974147
- [Background] Lindstedt S, Lindstedt G. Distribution and Excretion of Carnitine in the Rat. Acta. Chem. Scand. 1961;15:701-702
- [Background] Rebouche CJ, Engel AG. Carnitine metabolism and deficiency syndromes. Mayo Clin Proc. 1983 Aug;58(8):533-40. PMID 6348429
- [Background] Rebouche CJ, Paulson DJ. Carnitine metabolism and function in humans. Annu Rev Nutr. 1986;6:41-66. doi: 10.1146/annurev.nu.06.070186.000353. PMID 3524622
- [Background] Igarashi N, Sato T, Kyouya S. Secondary carnitine deficiency in handicapped patients receiving valproic acid and/or elemental diet. Acta Paediatr Jpn. 1990 Apr;32(2):139-45. doi: 10.1111/j.1442-200x.1990.tb00799.x. PMID 2143048
- [Background] Thurston JH, Hauhart RE. Amelioration of adverse effects of valproic acid on ketogenesis and liver coenzyme A metabolism by cotreatment with pantothenate and carnitine in developing mice: possible clinical significance. Pediatr Res. 1992 Apr;31(4 Pt 1):419-23. doi: 10.1203/00006450-199204000-00023. PMID 1570210
- [Background] Tein I, DiMauro S, Xie ZW, De Vivo DC. Valproic acid impairs carnitine uptake in cultured human skin fibroblasts. An in vitro model for the pathogenesis of valproic acid-associated carnitine deficiency. Pediatr Res. 1993 Sep;34(3):281-7. doi: 10.1203/00006450-199309000-00008. PMID 8134167
- [Background] Melegh B, Pap M, Morava E, Molnar D, Dani M, Kurucz J. Carnitine-dependent changes of metabolic fuel consumption during long-term treatment with valproic acid. J Pediatr. 1994 Aug;125(2):317-21. doi: 10.1016/s0022-3476(94)70218-7. PMID 8040784
- [Background] Tein I, Xie ZW. Reversal of valproic acid-associated impairment of carnitine uptake in cultured human skin fibroblasts. Biochem Biophys Res Commun. 1994 Oct 28;204(2):753-8. doi: 10.1006/bbrc.1994.2523. PMID 7980539
- [Background] Van Wouwe JP. Carnitine deficiency during valproic acid treatment. Int J Vitam Nutr Res. 1995;65(3):211-4. PMID 8830002
- [Background] Evangeliou A, Vlassopoulos D. Carnitine metabolism and deficit--when supplementation is necessary? Curr Pharm Biotechnol. 2003 Jun;4(3):211-9. doi: 10.2174/1389201033489829. PMID 12769764
- [Background] Coulter DL. Carnitine deficiency: a possible mechanism for valproate hepatotoxicity. Lancet. 1984 Mar 24;1(8378):689. doi: 10.1016/s0140-6736(84)92209-8. No abstract available. PMID 6142383
- [Background] Coulter DL. Carnitine, valproate, and toxicity. J Child Neurol. 1991 Jan;6(1):7-14. doi: 10.1177/088307389100600102. PMID 2002205
- [Background] Scriver C, Beautet A, Sly W, Valle D. The Metabolic Basis of Inherited Disease. New York: McGraw Hill, 1989
- [Background] Schaub J, Van Hoof F, Vis H. Inborn Errors of Metabolism. New York: Raven Press, 1991
- [Background] Standardization of Spirometry, 1994 Update. American Thoracic Society. Am J Respir Crit Care Med. 1995 Sep;152(3):1107-36. doi: 10.1164/ajrccm.152.3.7663792. No abstract available.
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831

RESULTS

PARTICIPANT FLOW:
Groups:
- SMA Type 1: All patients will receive VPA and carnitine.
  Valproic Acid and Levocarnitine: Drug: Valproic Acid and Levocarnitine; syrup; dosage is by weight
Period: Overall Study
Arm/Group | SMA Type 1
Started | 38
Completed | 25
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | SMA Type 1
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: months] | 5.52 (2.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 20
Region of Enrollment [Number; unit: participants]
  Canada | 2
  United States | 34
  Germany | 2

OUTCOME MEASURES:

1. Primary Outcome: Laboratory Safety Data
Time Frame: -2 weeks, + 2 weeks, 3 months, 6 months
Reporting Status: Not Posted

2. Primary Outcome: Anthropometric Measures of Nutritional Status (Body Mass Index [BMI] Z-scores, Weight for Length Ratios, Lean/Fat Mass Via DEXA, Growth Parameters, and Triceps Skinfold Measures)
Time Frame: -2 weeks, time 0, 3 months, 6 months
Population: 20 participants have baseline values, only 12 have 3 and 6 month values
Measure: Mean (Standard Deviation); unit: g
Arm/Group | SMA Type 1
Number analyzed (Participants) | 20
g
  Lean Mass Baseline | 4317.15 (1334.48)
  Lean Mass 3 months | 4993.92 (1676.13)
  Lean Mass 6 months | 5133.83 (2122.99)
  Fat Mass Baseline | 3011.37 (1467.83)
  Fat Mass 3 months | 3618.25 (1343.25)
  Fat Mass 6 months | 4316.08 (1857.16)

3. Secondary Outcome: Time to Death or Ventilator Dependence (Defined as >16 Hours/Day)
Time Frame: monthly
Reporting Status: Not Posted

4. Secondary Outcome: Primary Caregiver Functional Rating Scale for SMA Type I Subjects (PCFRS)
Time Frame: time 0, and monthly for 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Functional Motor Assessments: TIMPSI Scores
Time Frame: -2 weeks, time 0, 3 months, 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Quantitative SMN mRNA and Protein Measures
Time Frame: -2 weeks, time 0 , 3 months, or 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Maximum Ulnar CMAP Amplitude/Area and MUNE
Time Frame: -2 weeks, time 0, 3 months, 6 months
Reporting Status: Not Posted

8. Secondary Outcome: Whole Body DEXA Scanning for Lean Body Mass and Total Bone Mineral Density/ Content
Time Frame: -2 weeks or time 0, 3 months, 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | SMA Type 1
Serious Adverse Events (participants affected / at risk) | 29/38
Other Adverse Events (participants affected / at risk) | 36/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SMA Type 1 (N=38)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Congenital familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 7 (9)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 5 (6)
Bronchial Infection (Infections and infestations) | 1 (1)
Lip Infection (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 1 (2)
Wound Infection (Infections and infestations) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 13 (17)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SMA Type 1 (N=38)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Middle Ear Inflammation (Ear and labyrinth disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (3)
Fever (General disorders) | 12 (22)
Irritability (General disorders) | 2 (4)
Pain (General disorders) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 10 (12)
Allergic Reaction (Immune system disorders) | 1 (1)
Bronchial Infection (Infections and infestations) | 3 (3)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 5 (7)
Mucosal infection (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (2)
Skin Infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Weight Loss (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Nystagmus (Nervous system disorders) | 2 (2)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (15)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 12 (16)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No